CLINICAL TRIAL: NCT06841120
Title: Evaluation of Photobiomodulation Therapy with Diode Laser in Reversal of Maxillary and Mandibular Soft Tissue Local Anaesthesia in Paediatric Dentistry: Randomized Clinical Trial:a Randomized Clinical Trial
Brief Title: Reversal of Anaesthesia with Diode Laser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Recep Tayyip Erdogan University (Other)
Responsible Party: Principal Investigator, Ayça Kurt, Associate Professor, Recep Tayyip Erdogan University
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RecepTayyipErdoganUniversity
Record Dates: First submitted 2025-01-21; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-01

CONDITIONS: Photobiomodulation Therapy
Keywords: photobiomodulation therapy; diode laser; dental local anaesthesia; child

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Actual laser application (Experimental)
  Interventions: Device: Actual laser application
- Sham laser was applied symbolically (Sham Comparator)
  Interventions: Device: Sham laser application

INTERVENTIONS:
Device: Actual laser application — At approximately 45 minutes into the treatment session, subjects in the laser group received irradiation from a 4 W power, 810 nm diode laser (Fox; ARC Laser, GmbH, Nürnberg, Germany). The laser was operated in continuous mode, delivering 12-second shots per point using a therapy head with a point size of 0.38 cm². Each point received 6.3 J/cm² of laser energy, resulting in a total energy density of 37.8 J/cm² across 6 points.
  Arms: Actual laser application
Device: Sham laser application — Sham laser was applied symbolically as a diffused closed laser (targeted beam) at the same distance and simultaneously. Evaluations after laser irradiation were conducted by a responsible specialist physician who was not involved in performing the treatment procedures.
  Arms: Sham laser was applied symbolically

SUMMARY:
Background: After local anesthesia, which is frequently used in pediatric dentistry, long-term soft tissue numbness can cause various problems. The aim of this study was to evaluate the effectiveness of PBMT in reversing soft tissue anaesthesia in children following local anaesthesia administration.

Methods: In a split-mouth randomized study, 40 children aged 4 to 9 years, eligible to receive local infiltration injection on both maxillary (n=20) and mandibular (n=20) right and left sides, will included. Maxillary and mandibular quadrants will be randomly assigned to laser or sham laser groups. Normality will assessed using the Kolmogorov-Smirnov test. Categorical variables between laser and control groups will compared using the McNemar paired sample test. Significance will be set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* - Children whose parents signed the written informed consent form and who themselves gave assent,
* Children with a Frankl behaviour rating scale score of 3 or 4,
* Children aged between 4 and 9 years old who can understand soft tissue sensation and respond to it,
* Children requiring treatment with local infiltration anaesthesia for multiple teeth in both the mandible and maxilla,
* Children with no history of allergy to materials used for anaesthesia or sulphite,
* Children who have not taken any analgesic medication at least 24 hours before treatment,
* Children without any systemic conditions that would interfere with dental treatment under local anaesthesia.

Exclusion Criteria:

* Occurrence of an error during anaesthesia injection resulting in insufficient anaesthesia for treatment,
* Inability of the patient to provide clear assessments of response to soft tissue anaesthesia,
* Presence of systemic conditions that would prevent anaesthesia administration or dental treatment,
* Children requiring urgent dental treatment priority such as acute painful teeth.

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2023-01-18 (Actual); Primary Completion 2024-01-18 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Anesthesia reversal time | up to 30 minutes after procedure
  Until the first reversal of anesthesia, a palpation technique will be used to record every 10 minutes. With this technique, the presence of a sense of touch and tingling will be questioned. In order to obtain an objective answer, the child will be asked whether he/she knows what a tingling sensation is based on his/her previous experiences and will be told what and how this sensation is.

CONTACTS AND LOCATIONS:
Locations (1):
- Recep Tayyip Erdoğan University, Faculty of Dentistry, Rize, Rize Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No